CLINICAL TRIAL: NCT04926675
Title: Development of a Money Advice Intervention Within IAPT: Service User Case-studies
Brief Title: Development of a Money Advice Intervention Within IAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Professor Dame Til Wykes, Professor, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300734
Record Dates: First submitted 2021-05-28; First posted 2021-06-15 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Mental Health Issue; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Interventional study of adding money advice to psychological treatment compared to usual treatment from routine data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined intervention (Experimental): Participants accessing one-to-one psychological therapy from the IAPT service will be asked if they have any money worries affecting their mental health. Suitable participants will be offered one-to-one support from a money advisor, who they will access in tandem to their therapy.
  Interventions: Behavioral: Psychological Therapy; Behavioral: Debt Advice

INTERVENTIONS:
Behavioral: Psychological Therapy — Participants will be receiving their one-to-one psychological therapy from IAPT as usual. They typically receive between 6 and 12 sessions with a psychological practitioner.
Behavioral: Debt Advice — Participants will receive one-to-one support from a Citizen's Advice (CA) money advisor for as long as needed to resolve any money worries currently affecting their mental health.

SUMMARY:
This study is the second study of a larger project and will begin the process of testing and the development of an integrated intervention on a series of case studies. The combined intervention provides psychological therapy and debt advice in tandem. The treatment pathway is based on interviews and focus groups with service users and staff and the themes that emerged. It will be trialled in the NHS' Improving Access to Psychological Therapies (IAPT) service. Participants routinely accessing this service who have debt issues affecting their mental health will be asked if they'd like to also take up support for their money worries, which will be provided by Citizen's Advice (CA). Researchers will take exit interviews with both service users and staff at the end of the treatment to develop the protocol further. Researchers will also assess measures of mental health and wellbeing that are routinely taken by IAPT to review the intervention.

ELIGIBILITY:
Inclusion Criteria:

* IAPT clients referred for 'high-intensity' one-to-one treatment in the South London and Maudsley NHS Trust (SLaM)
* Have mental health problems and experience of money problems that are effecting these
* Can access technology

Exclusion Criteria:

* Inability to give informed consent due to mental incapacity (as assessed by IAPT therapists)
* Participants whose care team specify concerns regarding taking part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Reliable recovery - anxiety | 6-12 weeks
  Changes on the Generalized Anxiety Disorder - 7 (GAD-7), from above clinical cut off pre intervention (> 5) to below cut off post intervention (<5). The seven items on the scale ask participants to rate on a scale of 0 (not at all) to 3 (nearly everyday) how often they were bothered by each symptom. Total scores can range from 0 - 21, with higher scores indicating more anxiety.
Reliable recovery - depression | 6-12 weeks
  Patient Health Questionnaire - 9 (PHQ-9), from above clinical cut off pre intervention (> 5) to below cut off post intervention (<5). The nine items on the scale ask participants to rate on a scale of 0 (not at all) to 3 (nearly everyday) how often they were bothered by each symptom. Total scores can range from 0 - 27, with higher scores indicating more depressive symptoms.
Reliable recovery - adjustment | 6 - 12 weeks
  Work and Social Adjustment Scale - 5 (WSAS-5), from above clinical cut off pre intervention (> 10) to below cut off post intervention (<10). The five items on the scale ask participants to rate on a scale of 0 (not at all) to 8 (very severely) how much they feel they are impaired for each task. Total scores can range from 0 - 40, with higher scores indicating more impairment across work and social tasks.

SECONDARY OUTCOMES:
Financial Outcomes and service satisfaction | 6-12 weeks
  This survey has been adapted for the purposes of this study. It uses questions taken from the audit measure of service satisfaction used by Citizen's Advice. Participants are asked to rate on a scale of 1 (not at all) to 5 (a great deal) how much they experienced six possible effects from the combined intervention. Scores range from 6 to 30, with higher scores indicating more positive outcomes in relation to personal finances from the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Til Wykes, Prof. Dame., Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No